CLINICAL TRIAL: NCT06402812
Title: The Perceived Mismatch Between Dose Recommendations of PKI's and the Clinical Practice
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 18620
Record Dates: First submitted 2024-04-29; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regulators: Regulators
  Interventions: Other: Interview
- Proefssionals: Professionals
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — A qualitative research study will be conducted using semi-structured interviews. The target population includes regulators involved in the registration of PKIs and healthcare professionals who use PKIs in clinical practice. Participants will be recruited until a rich understanding of the subject is reached.

SUMMARY:
A qualitative research study will be conducted using semi-structured interviews. The target population includes regulators involved in the registration of PKIs and healthcare professionals who use PKIs in clinical practice. Participants will be recruited until a rich understanding of the subject is reached.

DETAILED DESCRIPTION:
* Background Protein kinase inhibitors (PKIs) are increasingly used as targeted therapy in the treatment of cancer. Currently, most PKIs are administered following the recommended dosage from the registered label based on pharmacokinetic and pharmacodynamic data, toxicity and tumor response as observed in clinical trials. Often, the recommended dose is selected based on the principle of the maximum tolerated dose (MTD). However due to pharmacokinetic and pharmacokinetic differences within patients, this registered flat starting dose often leads to toxicity. In addition, the fit and selected clinical trial patients are not always representative of the patients in clinical practice. This raises the question if the policy around dose development and recommendation is optimal. The objective of this study is therefore to increase patient safety, by exploring the perceptions of regulators and healthcare professionals on the perceived mismatch between the recommended dosage and the dose used in clinical practice for PKIs.
* Main research question What are the perceptions from regulators and healthcare professionals regarding the dosing recommendations for PKIs in clinical practice?
* Design (including population, confounders/outcomes) A qualitative research study will be conducted using semi-structured interviews. The target population includes regulators involved in the registration of PKIs and healthcare professionals who use PKIs in clinical practice. Participants will be recruited until a rich understanding of the subject is reached.
* Expected results This research aims to contribute to patient safety of PKIs in cancer treatment by exploring the opinions regarding the dosing recommendations at registration and their use in clinical practice from regulators and healthcare professionals. By gathering perceptions from important, preselected, stakeholders regarding dose regulations for PKIs, substantive knowledge will be gathered on the subject. This study will increase the knowledge base on the sufficiency of the standards for dose recommendations regarding PKIs and potentially aid in the generation of new policy recommendations.

ELIGIBILITY:
Inclusion Criteria:

- Regulators involved in the regulation of oncolytic products. Healthcare professionals who prescribe PKI's as a treatment for cancer in clinical practice (e.g. oncologists).

Exclusion Criteria:

* No exclusion criteria will be maintained.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Regulators and professionals
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Interview | 3 months
  Spoken words of participants will be gathered via interviews which have been conducted following an pre-set up interview guide.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Broekman, MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No